CLINICAL TRIAL: NCT06271564
Title: Effectiveness of Topical Magnetite Zinc Oxide Composite Nanoparticles in the Management of Oral Potentially Malignant Lesions (A Randomized Controlled Clinical Trial)
Brief Title: Effectiveness of Topical Magnetite Zinc Oxide Composite Nanoparticles in the Management of Oral Potentially Malignant Lesions
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nourhane Adel Abdel Halim Omara, Resident at Oral Medicine and Periodontology Department, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-Rec IM012415
Record Dates: First submitted 2024-02-12; First posted 2024-02-22 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Oral Potentially Malignant Lesions
Keywords: Oral Potentially Malignant Lesions; OPL; Nanoparticles; ZNO

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetite Zno Composite Nanoparticles (Experimental): 5% topical ZnO-Fe3O4 Magnetic Composite NPs gel applied 3 times per day for 6 weeks
  Interventions: Drug: Magnetite ZnO Composite Nanoparticles
- Topical Placebo Gel (Placebo Comparator): Topical Placebo Gel containing water, glycerin and Hydroxypropyl methylcellulose applied 3 times per day for 6 weeks
  Interventions: Drug: Topical Placebo Gel

INTERVENTIONS:
Drug: Magnetite ZnO Composite Nanoparticles — Magnetite ZnO-Fe3O4 conjugated NPs retained inherent selective property of ZnO and magnetic property of Fe3O4 NPs and showed preferential cytotoxicity towards breast cancer cell line MDA-MB-231, with no significant cytotoxicity towards noncancerous Mouse Fibroblast NIH 3T3 cell
  Arms: Magnetite Zno Composite Nanoparticles
Drug: Topical Placebo Gel — Topical placebo gel containing water, glycerin and Hydroxypropyl methylcellulose will be applied 3 times daily for 6 weeks as a positive control group
  Arms: Topical Placebo Gel

SUMMARY:
ZnO nanoparticles are now being widely researched for their anticancer properties. They show relatively high biocompatibility. They also show selective cytotoxicity against cancerous cells in in vitro condition compared with other nanoparticles. They can be further surface engineered to show increased selective cytotoxicity. The synthesis process of ZnO nanoparticles is relatively easy, with a wide variety of methods. Owing to these different methods of synthesis, their size and size distribution can be easily controlled. One of the novel methods of synthesis of ZnO is Magnetite ZnO-Fe3O4 Composite Nanoparticles.Magnetite ZnO-Fe3O4 conjugated NPs retained inherent selective property of ZnO and magnetic property of Fe3O4 NPs and showed preferential cytotoxicity towards breast cancer cell line MDA-MB-231, with no significant cytotoxicity towards noncancerous Mouse Fibroblast NIH 3T3 cell.

DETAILED DESCRIPTION:
Two interventions will be used; Magnetite ZnO-Fe3O4 Composite NPs extract and Placebo gel in custom made inert hydrophilic adhesive gel paste will be prepared in Nanotechnology engineering service in Egypt (Nano Gate), to enhance the adhesiveness of the two study interventions to oral mucosa.Group I (Test Group): Will include 15 patients with OPLs that will be treated with 5% topical ZnO-Fe3O4 Magnetic Composite NPs gel applied 3 times per day33 for 6 weeks9.

Group II (Positive Control Group):

Will include 15 patients with oral lichen planus lesions that will be treated with Topical Placebo Gel applied 3 times per day for 6 weeks.

The whole study period will be 18 weeks; 6 weeks as an active treatment period starting 1 week after the biopsy is taken then treatment discontinued for all groups and patients will be followed up for another 12 weeks in a treatment-free period.IV-Treatment efficacy evaluation A) Clinical efficacy assessment The assessment will be carried out at 0, 6 weeks and 18 weeks after starting the treatment protocol.

1-Imaging of the oral marker lesion Standardized photographs of the oral marker lesion for each patient will be taken with the same digital camera and setting, the surface area of the lesion will be outlined and measured using specific image software.

Histopathological analysis B-

The biopsy specimens for each patient will be taken at baseline and after 6 weeks of the treatment period and at 18 weeks for follow up then formalin-fixed and paraffin-embedded for:

ELIGIBILITY:
Inclusion Criteria:

* Both genders ranged from 25 to 60 years.
* Clinically confirmed OPMLs: the clinical picture of oral erythroplakia includes well-demarcated red discs with a smooth or granular surface, leukoplakia is classified into four clinical types: type I, a flat white patch or plaque without red components; type II, a flat white patch or plaque with red components; type III, a slightly raised or elevated white plaque; and type IV, a markedly raised or elevated white plaque.
* Histopathological confirmed OPMLs with low or moderate dysplasia

Exclusion Criteria:

* Presence of systemic conditions as serious active or recurrent infections, malignancy, diabetes mellitus, hypertension, or significant heart, liver, or renal diseases. Assessed using a medical questionnaire guided by Cornell Medical Index
* Smoking 6 weeks before the clinical trial
* Known hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation as mentioned in history.
* Pregnancy or breastfeeding.
* Histological diagnosis of severe, or invasive oral squamous cell carcinoma.
* Vulnerable groups (Handicapped, orphans or prisoners).
* Any lesion less than 1 cm in diameter.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in the clinical size in Low to Moderate Dysplastic OPLs using Magnetite ZnO-Fe3O4 Composite NPs using standardized photographs of the oral marker lesion for each patient | 6 weeks
  the surface area of the lesion will be outlined and measured using specific image software.

SECONDARY OUTCOMES:
Effect of Magnetite ZnO-Fe3O4 Composite NPs on the change of the degree of Dysplasia during histopathological examination using a biopsy | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ola Ezzatt, A.Professor, Study Director — Faculty of Dentistry-Ain shams university
Locations (1):
- Faculty of Dentistry Ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided